CLINICAL TRIAL: NCT00764608
Title: Study of the Human Skin Microbiome
Status: Withdrawn | Type: Observational
Why Stopped: No Participants enrolled, per PI discretion
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Principal Investigator, Randall Wolcott, Prinicipal Investigator, Southwest Regional Wound Care Center
Other Study IDs: 56-RW-012
Record Dates: First submitted 2008-09-30; First posted 2008-10-02 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2015-11

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The subjects' samples will be analyzed using DNA methods in order to identify the types of microbes present on the swabs. Other substances such as proteins, RNA, and other metabolites may also be analyzed. DNA or other molecular components of the sample will be extracted. Alternately, microbes in the sample can be cultured directly. The samples will be explored using molecular analyses. The backbone of the analyses will be shotgun metagenomic sequencing and 16S rDNA amplicon sequencing. The results of these analyses will be used to identify and describe the microbiome of the skin.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- No Treatment

SUMMARY:
Numerous organisms live on and in healthy human skin. This study seeks to survey the diversity of this complex ecosystem by collecting samples from approximately 1000 individuals in order to determine the type of organisms living on their skin.

DETAILED DESCRIPTION:
Subjects age 18 and above may be included in the study. It is the goal of the study to survey multiple skin locations of humans at multiple time points. The subjects' samples will be analyzed using DNA methods in order to identify the types of microbes present on the swabs. Other substances such as proteins, RNA, and other metabolites may also be analyzed. DNA or other molecular components of the sample will be extracted. Alternately, microbes in the sample can be cultured directly. The samples will be explored using molecular analyses. The backbone of the analyses will be shotgun metagenomic sequencing and 16S rDNA amplicon sequencing. The results of these analyses will be used to identify and describe the microbiome of the skin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years of age or older.
* Subjects must be able to consent for themselves.
* Must be willing to participate to a swab of the skin.

Exclusion Criteria:

* Subjects cannot be 17 years of age or younger.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: It is the goal of the study to survey multiple skin locations of humans at multiple time points
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Numerous organisms live on and in healthy human skin. This study seeks to survey the diversity of this complex ecosystem by collecting samples from approximately 1000 individuals in order to determine the type of organisms living on their skin. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Randall Wolcott, MD, Principal Investigator — Southwest Regional Wound Care Center
Locations (1):
- Southwest Regional Wound Care Center, Lubbock, Texas, United States